CLINICAL TRIAL: NCT06244407
Title: A Single Dose, Randomized, Open-label, Two-way Crossover Bioequivalence Study of Fixed-dose Combination of Vildagliptin and Metformin HCI 50/1000 mg FCT and Reference Product (Galvus Met®) in Healthy Thai Volunteers Under Fed Conditions
Brief Title: The Bioequivalence Study of Fixed-dose Combination of Vildagliptin and Metformin HCI 50/1000 mg FCT Under Fed Conditions
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: International Bio service (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: BE23-014
Record Dates: First submitted 2024-01-29; First posted 2024-02-06 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-01

CONDITIONS: Healthy Volunteer
Keywords: Vildagliptin and Metformin Hydrochloride 50/1000 mg FCT; Bioequivalence Study
MeSH Terms: interventions — Vildagliptin; Metformin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vildagliptin and Metformin Hydrochloride 50mg 1000 mg Film-coated tablet (Experimental): Participants first received Vildagliptin and metformin HCl 50/1000 mg 1 tablet (Test product) in a fasting state. After a washout period of 7 days, they then recieved Galvus Met® 1 tablet (Reference product) in a fed state.
  Interventions: Drug: Vildagliptin and Metformin Hydrochloride 50mg 1000 mg Film-coated Tablets
- Galvus Met® (Active Comparator): Participants first received Galvus Met® 1 tablet (Reference product) in a fed state. After a washout period of 7 days, they then recieved Vildagliptin and metformin HCl 50/1000 mg (Test product) in a fed state.
  Interventions: Drug: Vildagliptin and Metformin Hydrochloride 50mg 1000 mg Film-coated Tablets

INTERVENTIONS:
Drug: Vildagliptin and Metformin Hydrochloride 50mg 1000 mg Film-coated Tablets — Vildagliptin and Metformin Hydrochloride 50/1000 mg Film-coated Tablets
  Other Names: Vildagliptin and Metformin Hydrochloride 50/1000 mg Film-coated Tablets

SUMMARY:
To determine and compare the rate and extent of absorption of a test formulation with that of a reference innovator formulation when given as equal labeled dose in healthy subjects under fed conditions

DETAILED DESCRIPTION:
This study is conducted to investigate bioequivalence information which is required to ensure therapeutic equivalence of a test product and a reference product as well as to be considered as one aspect of product quality. Bioequivalence is defined as the absence of a significant difference in the rate and extent to which the active ingredient or active moiety in pharmaceutical equivalents or pharmaceutical alternatives becomes available at the site of drug action when administered at the same molar dose under similar conditions in an appropriately designed study.

The manufacturer needs to formulate a generic Fixed-dose Combination of Vildagliptin and Metformin HCI 50/1000 mg FCT. This study has been planned to evaluate the pharmacokinetics of this formulation and determine its bioequivalence with the reference product, Galvus Met®, at the same dose.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Thai male or female subjects between the ages of 18 to 55 years
2. Body mass index between 18.5 to 30.0 kg/m2
3. Normal laboratory values, including vital signs and physical examination, for all parameters in clinical laboratory tests at screening Any abnormalities from the normal or reference range will be carefully considered clinically relevant by the physician as individual cases, documented in study files prior to enrolling the subject in this study.
4. Non-pregnant woman (negative pregnancy test) and not currently breast feeding
5. Female subjects abstain from either hormonal methods of contraception (including oral or transdermal contraceptives, injectable progesterone, progestin subdermal implants, progesterone-releasing IUDs, postcoital contraceptive methods) or hormone replacement therapy for at least 28 days prior to check-in in Period 1. Injectable contraceptives e.g. Depo-Provera® will be discontinued at least 6 months prior to check-in in Period 1. Subjects agree to use acceptable non-hormonal contraceptive methods such as condom, diaphragm, foams, jellies, or abstinence for at least 14 days prior to check-in in Period 1 until 7 days after the end of study in Period 2. Female subjects of non-childbearing potential must meet at least one of the following criteria prior to check-in in Period 1:

   * Postmenopausal for at least 1 year
   * Surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy) at least 6 months
6. Male subjects who are willing or able to use effective contraceptive e.g. condom or abstinence after check-in in Period 1 until 7 days after the end of study in Period 2.
7. Have voluntarily given written informed consent (signed and dated) by the subject prior to participating in this study

Exclusion Criteria:

1. History of allergic reaction or hypersensitivity to vildagliptin or metformin HCl or to any of the excipients
2. History or evidence of clinically significant renal, hepatic, gastrointestinal, hematological (e.g. anemia), endocrine (e.g. hypo-/hyperthyroid, diabetes), pulmonary or respiratory (e.g. asthma), cardiovascular (e.g. hypo-/hypertension), psychiatric, neurologic (e.g. seizures), allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing) or any significant ongoing chronic medical illness
3. Have high risk for coronavirus infection based on risk assessment questionnaire or diagnosed as confirmed case of COVID-19
4. History about administration of COVID-19 vaccine within 30 days prior to check-in in each Period.
5. History or evidence of type 1 diabetes mellitus or lactic ketoacidosis or diabetic ketoacidosis
6. Have abnormality of glucose (FBS)
7. Investigation with blood sample shows fasting blood glucose level less than 70 mg/dl or more than 99 mg/dl at screening
8. History or evidence of acute pancreatitis
9. History or evidence of bullous pemphigoid or exfoliative skin lesion
10. History or evidence of acute pancreatitis
11. History of sensitivity to heparin or heparin-induced thrombocytopenia
12. History of problems with swallowing tablet or capsule
13. Any condition possibly affecting drug absorption e.g. gastrectomy, enterectomy, gastritis or duodenal or gastric ulceration other than appendectomy
14. History of diarrhea or vomiting within 24 hours prior to check-in in each period
15. History or evidence of drug addict or investigation with urine sample shows a positive test for drug of abuse (morphine, marijuana or methamphetamine) 16.12-lead ECG demonstrating QTc >450 msec, a QRS interval >120 msec or with an abnormality considered clinically significant at screening. If QTc exceeds 450 msec, or QRS exceeds 120 msec, the ECG will be repeated two more times and the average of the three QTc or QRS values will be used to determine the subject's eligibility.

17.Have eGFR (CKD-EPI) <30 mL/min/1.73 m2 based on serum creatinine results, at the screening laboratory test or during enrollment.

18.Abnormal liver function, ≥1.5 times of upper normal limit of reference range for ALT, AST or bilirubin levels at screening laboratory test

19.Investigation with blood sample shows positive test for HBsAg

20.History or evidence of habitual use of tobacco or nicotine containing products and cannot abstain for at least 48 hours prior to check-in in Period 1 and continued for entire duration of the study

21.History or evidence of alcoholism or harmful use of alcohol (less than 2 years) i.e., alcohol consumption of more than 14 standard drinks per week for men and 7 standard drinks per week for women (A standard drink is defined as 360 mL of beer or 150 mL of wine or 45 mL of 40% distilled spirits, such as rum, whisky, brandy, etc.)

22.History or evidence of alcohol consumption or alcohol-containing products and cannot abstain for at least 48 hours prior to check-in in Period 1 and continued for entire duration of the study or alcohol breath test shows positive result In case of alcohol breath test result represents the alcohol concentration range of 1

* 10 mg% BAC and the physician carefully considers that the value came from other reasons, not from the alcohol drinking behavior of subjects, the test will be repeated two times separately, not more than 10 minutes. The result of the last time should be used for subject's eligibility which must be 0 mg%BAC

  23.History or evidence of habitual consume of tea, coffee, xanthine or caffeine containing products and cannot abstain for at least 48 hours prior to check-in in Period 1 and continued for entire duration of the study

  24.Consume or drink juice of grapefruit or orange or pomelo or its supplement / containing products and cannot abstain for at least 7 days prior to check-in in Period 1 and continued for entire duration of the study 25.Use of prescription or nonprescription drugs (e.g. paracetamol, furosemide, nifedipine, iodinated contrast agents, ranolazine, vandetanib, dolutegravir, cimetidine, phenothiazines, thyroid products, phenytoin, nicotinic acid, isoniazid., antidiabetic drugs (e.g. glyburide), NSAIDs, corticosteroids, sympathomimetic drugs, diuretics, antihypertensive drugs, etc.), herbal medications or supplements (e.g. St. John's wort), vitamins or mineral (e.g. iron) or dietary supplements within 14 days prior to check-in in Period 1 and continued for entire duration of the study

  26.Participated in other clinical trials within 90 days prior to check-in in Period 1 (except for the subjects who drop out or withdrawn from the previous study prior to Period 1 dosing) or still participates in the clinical trial or participates in other clinical trials during enrollment in this study

  27.Blood donation or blood loss ≥ 1 unit (1 unit is equal to 350-450 mL of blood) within 90 days prior to check-in in Period 1 or during enrollment

  28.Subjects with poor venous access or intolerant to venipuncture

  29.Unwilling or unable to comply with schedule visit, treatment plan and other study procedures until end of study

  30.Inability to communicate well (i.e. language problem, poor mental development, psychiatric illness or poor cerebral function) that may impair the ability to provide written informed consent or cooperate with clinical team

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-05-23 (Estimated); Primary Completion 2024-05-25 (Estimated); Study Completion 2024-06-02 (Estimated)

PRIMARY OUTCOMES:
Plasma Area Under the Curve (AUC(0 to 36hr)) for Vildagliptin and Metformin | Through 36 Hours Post Dose]
  Plasma Area Under the Curve of Vildagliptin and Metformin

CONTACTS AND LOCATIONS:
Overall Officials: Uthai Suvanakoot, Ph.D.Pharm, Principal Investigator — International Bio service

IPD SHARING:
Plan to Share IPD: No
Confidential